CLINICAL TRIAL: NCT05822713
Title: Randomized, Double-blind, Placebo-controlled Phase III Study of Amisulpride for IV Injection as Prophylaxis Against Post-operative Nausea and Vomiting
Brief Title: A Comparison of the Efficacy of Amisulpride and Placebo in the Prevention of PONV in Patients at Moderate-to-high Risk of PONV.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qilu Pharmaceutical (Hainan) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: QLG2069-AMS-301
Record Dates: First submitted 2023-03-27; First posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-04

CONDITIONS: PONV
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Amisulpride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Amisulpride at 5mg was given by slow iv administration during1 to 2 min at induction of anesthesia
  Interventions: Drug: Amisulpride
- Placebo (Placebo Comparator): Placebo was given by slow iv administration during1 to 2 min at induction of anesthesia
  Interventions: Drug: Amisulpride Placebo

INTERVENTIONS:
Drug: Amisulpride — 5mg/2ml
  Arms: Experimental
Drug: Amisulpride Placebo — 2ml
  Arms: Placebo

SUMMARY:
A comparison of the efficacy of Amisulpride and placebo in the prevention of PONV in patients at moderate-to-high risk of PONV.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria:

1. Participant understand the study procedures and methods, voluntarily participate in this trial, and sign the informed consent.
2. Male or female patients ≥ 18 years of age and ≤75 years of age.
3. 18<BMI≤30kg/m^2，And weigh more than 45kg
4. Patients undergoing elective surgery(laparoscopic gynecological or abdominal surgery) under general anaesthesia requiring，and inhalation anesthesia is maintained for more than 1 hour, but patients who receive purely diagnostic surgery cannot be enrolled;
5. Patients with at least 2 of the following risk factors for PONV:

   Past history of PONV and/or motion sickness Habitual non-smoking status Female sex Expected to receive opioid analgesia post-operatively
6. American Society of Anesthesiologists (ASA) risk score I-III -

Exclusion Criteria:

1. Patients undergoing day case surgery
2. Patients undergoing intra-thoracic, transplant or central nervous system surgery or any surgery where post-operative emesis may pose a significant danger to the patient
3. Patients planned to receive only a local anaesthetic and/or regional neuraxial (intrathecal or epidural) block
4. Patients who are scheduled to be transferred to the ICU after surgery;
5. Patients who are expected to need a naso- or oral-gastric tube in situ after surgery is completed
6. Patients who have a documented, clinically significant cardiac arrhythmia or congenital long QT syndrome（Male≥ 450 ms female≥ 460ms）.
7. Adequate hepatic and renal function, Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2.5 x upper limit normal (ULN)，Bilirubin ≥ 1.5 x ULN，Creatinine ≥ 1.5x ULN
8. Patients who have received Amisulpride active ingredient for any indication within the last 2 weeks
9. Patients who are allergic to Amisulpride active ingredient or any of the excipients of Amisulpride
10. Patients with a significant, ongoing history of vestibular disease or dizziness
11. Intestinal obstruction
12. Patients with a known prolactin-dependent tumour (e.g. pituitary gland prolactinoma or breast cancer) or phaeochromocytoma.
13. Patients with pre-existing nausea or vomiting in the 24 hours before surgery
14. Patients treated with regular anti-emetic therapy including corticosteroids
15. Patients being treated with medications which could induce torsades de pointes, including Class Ia antiarrhythmic agents such as quinidine, disopyramide, procainamide; Class III antiarrhythmic agents such as amiodarone and sotalol; and other medications such as bepridil, cisapride, thioridazine, methadone, IV erythromycin, IV vincamine, halofantrine, pentamidine, sparfloxacin
16. Patients being treated with levodopa or other dopamine drugs
17. Patients who are pregnant or breast feeding.
18. Participant who has a history of drug or alcohol abuse within 6 months before randomization
19. Patients diagnosed with Parkinson's disease ，Patients with a history of epilepsy.
20. Patients who have received anti-cancer chemotherapy in the previous 4 weeks of surgery
21. Patients who have participated in other clinical research trials within 3 months before randomization
22. Participant who may increase study-related risks or interfere with the interpretation of study results in the opinion of the investigator, who are considered unsuitable for enrollment by the investigator and/or the sponsor.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 516 (Estimated)
Dates: Start 2023-04-29 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint was the composite measure complete response | 24 hours after the end of surgery
  defined as no episodes of emesis (vomiting or retching) and no use of rescue medication in the first 24h after wound closure

SECONDARY OUTCOMES:
Incidence of no Nausea | 24 hours after end of surgery
  Count of patients experiencing an episode of no nausea scored < 1 of 0-10 verbal response scale during the 24 hours period after the completion of surgery
Incidence of moderate and severe Nausea | 24 hours after end of surgery
  Count of participants with nausea score > 4 on 0-10 verbal response scale
Incidence of Emesis (Vomiting/Retching) | 24 hours after end of surgery
  An assessment of a participant experiencing an episode of emesis (vomiting/ retching) during the 24hours after the completion of the surgery
Use of Rescue Medication | 24 hours after end of surgery
Time to First Violation of Criteria for PONV | 24 hours after end of surgery
  Criteria for PONV are any episode of emesis or use of rescue medication in the 24 hours after the end of surgery

CONTACTS AND LOCATIONS:
Overall Officials: yi feng, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No